CLINICAL TRIAL: NCT02628912
Title: Pilot Study of Cardiopulmonary Fitness in Long-Term Survivors of HPV-related Oropharynx Cancers
Brief Title: Cardiopulmonary Fitness in Long-Term Survivors of HPV-related Oropharynx Cancers
Status: Withdrawn | Type: Observational
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 15-277
Record Dates: First submitted 2015-12-08; First posted 2015-12-11 (Estimated); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Oropharynx Cancers
Keywords: Cardiopulmonary Fitness; Long-Term Survivors; 15-277; HPV; Survivors
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Blood Specimen Collection; Exercise Test; Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood

GROUPS / COHORTS (1):
- long-term survivors of HPV-related oropharyngeal cancer: This is a cross-sectional pilot study of long-term survivors of HPV-related oropharyngeal cancer treated with CTRT who are at least three years from treatment completion. This study consists of a onetime assessment of cardiopulmonary fitness, physical function status, measurement of lean body mass, endothelial function quality of life assessment, medical history and blood laboratory evaluation for traditional cardiac risk factors, endocrine derangement and inflammation.
  Interventions: Other: blood draw; Behavioral: study questionnaire; Other: cardiopulmonary exercise testing (CPET); Other: DXA (dual-energy x-ray absorptiometry) scan

INTERVENTIONS:
Other: blood draw
Behavioral: study questionnaire
Other: cardiopulmonary exercise testing (CPET)
Other: DXA (dual-energy x-ray absorptiometry) scan

SUMMARY:
This study is being done to learn about how the participants lungs and heart are working after treatment for throat cancer. The investigators are looking to see if there is a long-term impact on overall health from the cancer treatment. The long-term goal of this study is to compare the participants overall quality of life to similarly aged people who have not had throat cancer.

DETAILED DESCRIPTION:
The goal of this study is not to test the impact of a specific intervention, but rather to evaluate the long-term cardiovascular health and quality of life of oropharyngeal cancer survivors using validated survey instruments, cardiopulmonary testing, and measurements of cardiac risk factors. Thus, no intervention, other than the assessments will be administered as part of the protocol. All participants will have received treatment according to the standard of care or a therapeutic clinical trial in which they may have participated previously. We will collect information about prior treatment from the electronic medical record (EMR).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosis of HPV+ squamous cell carcinoma of the oropharynx confirmed by the pathology department of MSKCC. Positive HPV status defined as chromogenic in situ hybridization with wide spectrum HPV probe (HPV III family 16 probe (Ventana) with affinity to HPV genotypes 16, 18, 31, 33, 35, 45, 51, 52, 56, 58, and
* 66) or p16 immunohistochemistry done in a Clinically Laboratory Improvement Amendment (CLIA) approved laboratory; if either of these 2 tests are positive, the patient is classified as HPV positive]
* Completed last treatment for oropharyngeal cancer (surgery, chemotherapy, or radiation) at least 3 years before enrollment in study
* Able to speak and read English
* Clinically shows no evidence of disease (NED)
* Received radiation therapy with a dose of at least 60Gy, at MSKCC as part of concurrent treatment
* Medical clearance from a member of the patient's healthcare team indicating no relative contraindications to undergoing a cardiopulmonary exercise test

Exclusion Criteria:

* Diagnosis with recurrent disease following completion of primary curative treatment
* History of any cancer other than HPV+ oropharyngeal squamous cell carcinoma, or current diagnosis of another cancer
* Current diagnosis of any of the following: Acute myocardial Infarction (within 3-5 days of any planned study procedures); Unstable angina; Arrhythmia; Syncope; Active endocarditis; Acute myocarditis or pericarditis; Symptomatic severe aortic stenosis; Heart failure; Acute pulmonary embolus or pulmonary infarction; Thrombosis of lower extremities; Suspected dissecting aneurysm; Pulmonary edema; Room air desaturation at rest ≤85%; Respiratory failure; Any acute non-cardiopulmonary disorders that may affect exercise performance or be aggravated by exercise (i.e., infection, renal failure, thyrotoxicosis); COPD or asthma noted in patients EMR.
* Mental impairment leading to an inability to cooperate or consent to this research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In protocol 10-111 "Surviving Oropharynx Cancer: Long-term Impact of Human Papillomavirus (HPV) on quality of life", a population of HPV+ oropharyngeal cancer survivors was identified. There are nearly 150 participants who have completed the one-time questionnaire on 10-111 who may meet the eligibility criteria for this study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
change in VO2peak | 1 year
  using cardiopulmonary exercise testing

CONTACTS AND LOCATIONS:
Overall Officials: Shrujal Baxi, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/